CLINICAL TRIAL: NCT03684122
Title: A Safety and Efficacy Study of the Effects of Mesenchymal Stem Cells (MSCs) Differentiated Into Neural Stem Cells (NSCs) on the Motor and Non-motor Symptoms in People With Parkinson's Disease (PD).
Brief Title: Use of Mesenchymal Stem Cells (MSCs) Differentiated Into Neural Stem Cells (NSCs) in People With Parkinson's (PD).
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Fatima Jamali, Head of Neuroscience Research, University of Jordan
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PKUJCTC
Record Dates: First submitted 2018-09-23; First posted 2018-09-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Parkinson Disease
Keywords: Umbilical cord Mesenchymal Stem Cells; Parkinson Disease; Neurodegenerative; allogeneic
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Injection of Umbilical cord derived MSCs (Experimental): Allogenic Umbilical Cord derived stem cells injected intravenously to enrolled PD patients
  Interventions: Biological: Injection of Umbilical cord derived MSCs
- Injection of MSCs differentiated into neural stem cells NSCs (Experimental): Allogenic Umbilical Cord derived stem cells (MSCs) differentiated into neural stem cells (NSCs) injected intrathecaly and intravenously to enrolled PD patients.
  Interventions: Biological: Injection of Umbilical cord derived MSCs

INTERVENTIONS:
Biological: Injection of Umbilical cord derived MSCs — Allogenic umbilical cord derived MSCs which are to be injected intrathecally and intravenously as a treatment option for consenting PD patients
  Other Names: injection of Umbilical cord derived MSCs differentiated into neural stem cells NSCs.

SUMMARY:
This study aims to examine the short term and long term safety outcomes of the treatment of PD patients with umbilical cord derived stem cells as indicated by the presence of adverse events that are confirmed to be related to the therapy.

DETAILED DESCRIPTION:
This study is predicted to confirm the safety of the use of allogeneic mesenchymal stem cell (MSCs) differentiated into neural stem cells (NSCs) in one of the most common neurological diseases. It will also aid in the better understanding of the role of stem cell therapy in relation to motor and non-motor symptoms in people with Parkinson disease. The safety outcomes would encourage launching similar larger studies. And also to facilitate the treatment and outcome results by giving differentiated mesenchymal stem cells (MSCs) into neural stem cells (NSCs) rather than allow the cells to differentiate inside the body. While the efficacy results if encouraging, would mean an improvement in the disability associated with PD and reduction in the life-time care and treatment provided to this category of patients in Jordan and the Arab region.

ELIGIBILITY:
Inclusion Criteria:

* Non- smokers
* Diagnosis of PD between 1 to 7 years
* Robust response to dopaminergic therapy (defined as greater than 33% reduction in symptoms (on the Unified Parkinson's Disease Rating Scale; UPDRS) when measured in the ON medicine state compared to OFF state.
* If subject is taking any central nervous system acting medications (e.g., benzodiazepines, antidepressants, hypnotics) regimen must be optimized and stable for 90 days prior to the screening visit.
* A stable Parkinson's disease symptomatic therapy for at least 90 days prior to screening and not projected to require additional Parkinson's disease symptomatic therapy for at least one year from the baseline visit.
* Women of childbearing potential will be required to use a reliable form of contraception from 30 days prior to baseline visit until 6 months after treatment
* A clear infectious panel examination including Hepatitis B, C, Human immunodeficiency virus (HIV), Syphilis

Exclusion Criteria:

* Atypical or drug-induced Parkinsonism.
* A UPDRS rest tremor score of 3 or greater for any limb on medication
* A Montreal Cognitive Assessment (MoCA) score of less than 25.
* Clinical features of psychosis or refractory hallucinations.
* Uncontrolled seizure disorder, defined as a seizure within the last 6 months.
* Developmental delay.
* Hepatic disease or altered liver function as defined by alanine transaminase (ALT) >150 U/L and or T. Bilirubin >1.6 mg/dl at admission.
* Presence of clinically refractory orthostatic hypotension at the screening or baseline visit defined as greater than or equal to 20 mmHg change in systolic Blood pressure (BP) and greater than or equal to 10 mmHg change in diastolic BP from sitting position to standing after 2 minutes that does not respond to medical treatment or baseline sitting BP less than 90/60.
* History of congestive heart failure, clinically significant bradycardia, presence of 2nd or 3rd degree atrioventricular block.
* Active malignancy or diagnosis of malignancy within 5 years prior to the start of screening (Cancer free for at least 5 years is permitted; skin cancers, except for melanoma, are permitted).
* History of strokes or traumatic brain injury.
* Major surgery within the previous 3 months or planned in the ensuing 6 months.
* Clinically significant abnormalities in the Screening Visit laboratory studies.
* History of use of an investigational drug within 30 days prior to the screening visit.
* History of brain surgery for PD.
* Unable to return for follow-up visits for clinical evaluation, laboratory studies, or imaging evaluation.
* Any other condition that the investigator feels would pose a significant hazard to the patient if enrolled or complicate the study assessments.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2021-09-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]) as a result of the injection | 6 months
  Side effects will be reported as Incidence of treatment-emergent adverse events (TEAEs), serious TEAEs, related TEAEs, severe TEAEs

SECONDARY OUTCOMES:
Drug Reduction Rate test | 6 months
  Based on reduction rate, the efficacy can be defined as complete remission, partial remission, effective and invalid. The reduction rate will be 100%, >50%, >25%-50%, ≤25% for complete remission, partial remission, effective and invalid.
Tractography | 6 months
  Gait and balance analysis system.
Blood-based biomarkers | 6 months
  Blood-based biomarkers will be analysed which include the concentration in ng/ul of α-synuclein, uric acid, epidermal growth factor, apolipoprotein-A1, and peripheral inflammatory markers using the 20-plex Luminex technology.
Cerebrospinal Fluid (CSF) based biomarkers | 6 months
  Cerebrospinal Fluid (CSF) based biomarkers such as α-synuclein (αSyn), β-amyloid 1-42 (Aβ42), tau,phosphorylated tau, and neurofilament light chain will be analyzed and their concentration were measured in ng/ul.

CONTACTS AND LOCATIONS:
Overall Officials: Abdallah Awidi, MD, Study Director — Cell Therapy Center
Locations (1):
- Cell Therapy Center, University of Jordan, Amman, Jordan

REFERENCES:
- [Derived] Jamali F, Aldughmi M, Khasawneh MW, Dahbour S, Salameh AA, Awidi A. A New Tool for Safety Evaluation and a Combination of Measures for Efficacy Assessment of Cotransplanting Human Allogenic Neuronal Stem Cells and Mesenchymal Stem Cells for the Treatment of Parkinson Disease: Protocol for an Interventional Study. JMIR Res Protoc. 2021 Oct 22;10(10):e29695. doi: 10.2196/29695. PMID 34677138